CLINICAL TRIAL: NCT00373711
Title: Comparison of I-124 PET/CT, F-18 FDG PET/CT and I-123 Whole Body Scintigraphy for Recurrent Thyroid Cancer Detection
Brief Title: Comparison of I-124 PET/CT, F-18 FDG PET/CT & I-123 Whole Body Scintigraphy for Recurrent Thyroid CA
Status: Withdrawn | Type: Observational
Why Stopped: Abandoned
Sponsor: Stanford University (Other)
Responsible Party: Iain Ross McDougall, Stanford University School of Medicine
Other Study IDs: END0003; 97454 (Other: Stanford University Alternate IRB Approval Number); END0003 (Other: Stanford University)
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2011-04

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Iodine-124; Iodine-123; Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Iodine-124 — 2 mCi, oral
  Other Names: Eastern Isotopes
Drug: Iodine-123 — 2 mCi, oral
  Other Names: MDS Nordion
Drug: F-18 FDG — 10-15 mCi, iv
  Other Names: Fludeoxyglucose (18 F); fluorodeoxyglucose (18 F); MIPS

SUMMARY:
The management of thyroid cancer patients with suspicion of recurrent disease based on rising/detectable levels of thyroglobulin (Tg) involves imaging with iodine-123 whole body scintigraphy (I-123 WBS) and F-18 FDG PET/CT. However, the disease is not always detected. The use of another iodine isotope (I-124) with positron emitting characteristics for PET/CT may allow better identification of recurrent disease, thus allowing for more patients to be treated with I-131 as a curative attempt.

DETAILED DESCRIPTION:
The management of thyroid cancer patients with suspicion of recurrent disease based on rising/detectable levels of thyroglobulin (Tg) involves imaging with iodine-123 whole body scintigraphy (I-123 WBS) and F-18 FDG PET/CT. However, the disease is not always detected. The use of another iodine isotope (I-124) with positron emitting characteristics for PET/CT may allow better identification of recurrent disease, thus allowing for more patients to be treated with I-131 as a curative attempt.

Conducting this study we hope to find whether I-124 PET/CT allows for detection of more lesions in patients with suspected recurrent thyroid cancer than the current standard of care represented by I-123 WBS and F-18 FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:- Patient at Nuclear Medicine clinic at Stanford University Medical Center

* Treated thyroid cancer.
* Detectable levels of Tg.
* Referred for I-123 WBS and F-18 FDG PET/CT for detection of recurrent thyroid cancer.
* Able to have a I-124 PET/CT the day after I-123 WBS and F-18 FDG PET/CT
* Patients older than 18-year-old.
* Patients with history of treated thyroid cancer and suspected recurrent thyroid cancer based on detectable levels of Tg.
* Patients must have I-123 WBS and F-18 FDG PET/CT performed prior to the I-124 PET/CT.
* Patients must understand and voluntarily sign an Informed Consent form after the contents have been fully explained to them. Exclusion Criteria:- Patients who are not eligible for I-123 WBS and F-18 FDG PET/CT.
* Patients who cannot complete I-123 WBS and F-18 FDG PET/CT.
* Pregnant women.
* Healthy volunteers.
* Patients participating in other research studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Thyroid cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford University; Iain Ross McDougall, Principal Investigator — Stanford University